CLINICAL TRIAL: NCT07286266
Title: A Randomized, Open-label, Multicenter, Phase 3 Study to Investigate GSK5733584 Compared With Chemotherapy in Participants With Platinum-resistant Ovarian Cancer
Brief Title: A Study to Investigate GSK5733584 Compared With Chemotherapy in Participants With Platinum-resistant Ovarian Cancer (BEHOLD-Ovarian01)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 224031; 2025-523361-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-12; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Neoplasms
Keywords: Platinum-resistant Ovarian Cancer; GSK5733584; Paclitaxel; Pegylated liposomal doxorubicin (PLD); Topotecan; Gemcitabine; Antibody-drug conjugate; BEHOLD-Ovarian01
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; liposomal doxorubicin; Topotecan; Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The independent central reviewer assessing primary outcome data will be masked (blinded) from participants treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK5733584 (Experimental): Participants will receive GSK5733584
  Interventions: Drug: GSK5733584
- Standard of care (Active Comparator): Participants will receive standard of care chemotherapy (Paclitaxel or PLD or Topotecan or Gemcitabine) as per investigator's choice
  Interventions: Drug: Paclitaxel; Drug: Pegylated liposomal doxorubicin (PLD); Drug: Topotecan; Drug: Gemcitabine

INTERVENTIONS:
Drug: GSK5733584 — GSK5733584 will be administered
  Arms: GSK5733584
Drug: Paclitaxel — Paclitaxel will be administered
  Arms: Standard of care
Drug: Pegylated liposomal doxorubicin (PLD) — PLD will be administered
  Arms: Standard of care
Drug: Topotecan — Topotecan will be administered
  Arms: Standard of care
Drug: Gemcitabine — Gemcitabine will be administered
  Arms: Standard of care

SUMMARY:
This study specifically aims to evaluate how well GSK5733584 works in treating ovarian cancer compared to standard treatments. The study also assesses whether GSK5733584 is safe and tolerated well by participants compared to standard treatments and aims to provide a better understanding of the main side effects of the drug.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the legal age of consent in the jurisdiction in which the study is taking place at the time of signing the Informed Consent Form (ICF).
* Has epithelial ovarian, primary peritoneal or fallopian-tube cancer with a histologically confirmed diagnosis of high grade serous, high grade endometrioid, or clear cell carcinoma, or carcinosarcoma that is resistant to platinum-based therapy.

Platinum-resistance is defined as follows:

* Participants who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum therapy, must have had a response (CR, PR, stable disease) and then progressed from >3 months to ≤6 months after the last dose of platinum therapy.
* Participants who have received >1 line of platinum therapy must have progressed on or ≤6 months after the date of the last dose of platinum therapy.

  • Has received at least 1 but no more than 3 prior lines of systemic anti-cancer therapy, and for whom single-agent therapy is appropriate as the next line of treatment. Participants who received mirvetuximab soravtansine as prior therapy are permitted to have received up to 4 prior lines. Prior lines of therapy are defined as follows:
* Adjuvant ± neoadjuvant are considered one line of therapy.
* Maintenance therapy (e.g., bevacizumab, [Poly adenosine diphosphate-ribosylation (ADP) ribose polymerase inhibitor (PARPi)] will be considered as part of the preceding line of therapy (i.e., not counted independently).
* Therapy changed to another agent in the same class due to toxicity in the absence of progression will be considered as part of the same line (i.e., not counted independently).
* Unplanned addition or switching to a new drug in a different class is considered a separate line of therapy.
* Hormonal therapy will be counted as a separate line of therapy unless it was given as maintenance.

  * Has received prior treatment with Mirvetuximab soravtansine (MIRV), bevacizumab and/or PARPi if the participant was considered a candidate for this treatment and the treatment is locally available.
  * Has at least one Target lesion (TL) per RECIST 1.1, as determined by the investigator. Measurable lesions that have been previously irradiated and have been shown to be progressing following irradiation may be considered as TLs.
  * Has provided a Formalin fixed, paraffin embedded (FFPE) tumor tissue sample sufficient for the central assessment of B7 homolog 4 protein (B7-H4) expression, with the result of B7-H4 expression testing available prior to date of randomization.
  * Is eligible to receive 1 of the standard of care interventions if randomized to physician's choice arm. Participants not selected to receive taxane as physician's choice regimen must have previously received taxane-based treatment in the platinum-resistant setting or be intolerant to taxane-based treatment.
  * A female participant is eligible to participate if they are not pregnant or breastfeeding, and one of the following conditions applies:
* Is a Participant of non-childbearing potential (PONCBP) OR
* Is a Participant of childbearing potential (POCBP) and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, 30 days prior to Cycle 1 Day 1 (C1D1) and during the study intervention period and for at least 8 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.

  • A POCBP must have a negative, highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention
* If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

  * Is capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the ICF and in the study protocol.
  * Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Has adequate organ function

Exclusion Criteria:

* Has primary platinum-refractory Ovarian Cancer (OC), defined as disease that did not respond to or has progressed within <3 months of the final dose of first line platinum containing chemotherapy.
* Has a malignancy (except disease under study) that has progressed or required active treatment within 36 months prior to date of randomization, except for basal cell or squamous cell carcinomas of the skin, in-situ carcinomas (e.g., breast, cervix, bladder) that have been resected with no evidence of metastatic disease, or that is otherwise considered cured by the investigator.
* Has known sensitivity to study intervention components or excipients or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.
* Has untreated brain or CNS metastases or brain/CNS metastases that have progressed (e.g., evidence of new or enlarging brain metastasis or new neurologic symptoms attributable to brain/CNS metastases). Participants with previously treated and clinically stable brain/CNS metastases and who have completed all corticosteroid therapy for ≥14 days prior to date of C1D1 are not excluded from participation.
* Has any evidence of current ILD or pneumonitis, or a prior history of ILD or non-infectious pneumonitis.
* Has ongoing adverse reaction(s) from prior therapy that has (have) not recovered to ≤Grade 1 or to the baseline status preceding prior therapy, excluding e.g., alopecia, hearing loss, vitiligo, endocrinopathy managed with replacement therapy, and Grade 2 neuropathy, or that the investigator, with the agreement of the sponsor, considers to be not clinically relevant for the tolerability of study intervention in the current clinical study.
* Has any serious and/or unstable medical or psychiatric disorder or other condition(s) (including laboratory assessment abnormalities) that could interfere with the participant's safety, obtainment of informed consent, or compliance to the study procedures, including requirements for the Follow-up Period of the study.
* Has had any major surgery within 28 days prior to date of C1D1 or received focal radiotherapy within 21 days prior to date of C1D1.
* Has received treatment with an investigational agent within 30 days prior to date of C1D1.
* Has received treatment with any cytotoxic chemotherapy drugs or other anti-tumor drugs (including endocrine therapy, molecular targeted therapy, immunotherapy, biotherapy, or investigational agent) within 30 days or 5 half-lives, whichever is shorter, prior to date of C1D1; or need to continue these drugs during study participation.
* Has ever received prior therapy with topoisomerase I inhibitors (e.g., topotecan) or ADC with a topo1i payload, or B7-H4 targeted therapy.
* Has received any live vaccine within 30 days prior to date of C1D1.
* Has received treatment with strong or moderate inhibitor of Cytochrome P450 3A4 (CYP3A4) or Cytochrome P450 2D6 (CYP2D6), strong or moderate inducer of CYP3A4, inhibitor of P-glycoprotein (P-gp) or Breast cancer resistant protein (BCRP), or inducer of P-gp within 14 days prior to date of C1D1 or anticipates their use during study participation and up to 30 days after the last dose of study intervention administration.
* Use of drugs known to prolong the QT interval or potentially cause torsades de pointes; or need to continue these medications during the study and up to 30 days after the last dose of study intervention.
* Has received any transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including Granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 14 days prior to date of C1D1.
* For participants receiving PLD only: Has baseline Left ventricular ejection fraction (LVEF) <50% or lower than institutional lower limits of normal.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 450 (Estimated)
Dates: Start 2026-03-03 (Estimated); Primary Completion 2030-01-16 (Estimated); Study Completion 2030-01-16 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by BICR | Up to approximately 202 weeks
  PFS is defined as the time from the date of randomization to the date of first documented Progressive Disease per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) by Blinded independent central review (BICR) assessment or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 202 weeks
  OS is defined as the time from the date of randomization to the date of death due to any cause

SECONDARY OUTCOMES:
PFS by investigator assessment | Up to approximately 202 weeks
  PFS is defined as the time from the date of randomization to the date of first documented PD per RECIST 1.1 by investigator assessment or death from any cause, whichever occurs first
Objective response rate (ORR) by BICR | Up to approximately 202 weeks
  ORR is defined as the percentage of participants with best overall response of either complete response (CR) or partial response (PR) per RECIST 1.1 by BICR assessment
Duration of Response (DOR) by BICR | Up to approximately 202 weeks
  DOR is defined as the time from the date of first documented objective response (CR or PR) per RECIST 1.1 by BICR assessment to the date of first documented Progressive Disease (PD) per RECIST 1.1 by BICR assessment or death due to any cause, whichever occurs first
ORR by investigator assessment | Up to approximately 202 weeks
  ORR is defined as the percentage of participants with best overall response of either CR or PR per RECIST 1.1 by investigator assessment
DOR by investigator assessment | Up to approximately 202 weeks
  DOR is defined as the time from the date of first documented objective response (CR or PR) per RECIST 1.1 by investigator assessment to the date of first documented PD per RECIST 1.1 by investigator assessment or death due to any cause, whichever occurs first
PFS2 | Up to approximately 202 weeks
  PFS2 is defined as the time from the date of randomization to the date of first documented investigator-assessed clinical or radiographical progression following the first subsequent anticancer therapy and after the progression event used for PFS, or death from any cause, whichever occurs first
Number of participants with Treatment-emergent adverse event (TEAEs), Adverse event of special interest (AESIs) and Treatment-emergent serious adverse event (TESAEs) | Up to approximately 202 weeks
Number of participants with TEAEs/AESI/TESAEs leading to dose modifications or study intervention discontinuation | Up to approximately 202 weeks
Number of participants with changes in vital signs, laboratory tests (hematology and clinical chemistry), and Electrocardiogram (ECG) | Up to approximately 202 weeks
Serum concentration of GSK5733584 (conjugated antibody and payload) | Up to approximately 202 weeks
Number of participants with Antidrug antibody (ADA) and Neutralizing Antibody (NAb) against GSK5733584 | Up to approximately 202 weeks
Titers of ADA against GSK5733584 | Up to approximately 202 weeks
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) score | Up to approximately 202 weeks
  The EORTC QLQ-C30 includes 30-item questionnaire for evaluating the health-related quality of life (HRQoL) of participants participating in cancer clinical studies. The following domains will be measured: Global health status (GHS)/ Quality of Life (QoL), physical functioning, role functioning Participants responses on these items are . averaged and then transformed to scores . ranging from 0 to 100. Higher . score indicates better functioning or a better . overall state of health.
Change from baseline in EORTC QLQ-Ovarian Cancer Module (OV28) score | Up to approximately 202 weeks
  The EORTC QLQ-OV28 includes a 28-item questionnaire for evaluating ovarian cancer-specific symptoms and concerns in participants of cancer clinical studies. These include items that assess symptoms in the abdominal/gastrointestinal domain. Scores are averaged and transformed to a 0 to 100 scale; higher scores indicate a greater symptom burden, while lower scores reflect fewer symptoms.
Time to deterioration (TTD) of EORTC QLQ-OV28 | Up to approximately 202 weeks
  TTD is defined as the time from the date of randomization to the first confirmed clinically meaningful deterioration on the abdominal/gastrointestinal symptom domain of the EORTC QLQ-OV28
TTD of EORTC QLQ-C30 | Up to approximately 202 weeks
  TTD is defined as the time from the date of randomization to the first confirmed clinically meaningful deterioration on any of the following EORTC QLQ-C30 domains: physical functioning, role functioning and Global Health Status (GHS)/ Quality of Life (QoL).
Maximum Post-baseline Patient-reported outcome Common Terminology Criteria for Adverse Events (PRO-CTCAE) Score | Up to approximately 202 weeks
  The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicities in participants in cancer clinical trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE. A subset of items selected from the PRO-CTCAE item library will be assessed. This measure captures maximum post-baseline PRO-CTCAE score for each frequency, severity and/or interference of symptomatic AEs
Change from baseline in CA-125 tumor marker [units per milliliter (U/mL)] | Up to approximately 202 weeks

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf